CLINICAL TRIAL: NCT03231241
Title: SunStar Project to Explore the Chronification Process in Headache Through Functional Imaging, Deep Phenotyping, and Analysis of CSF of Blood Products
Brief Title: Analysis of Headache Chronification With Imaging, Deep Phenotyping, and Proteomics
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Cowan, Director and Chief, Division of Headache Medicine, Stanford University
Other Study IDs: SunStar
Record Dates: First submitted 2017-07-14; First posted 2017-07-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-12

CONDITIONS: Chronic Daily Headache; Chronic Migraine
Keywords: Headaches; Tension-Type Headache; New Daily Persistent Headache (NDPH); Migraine
MeSH Terms: conditions — Headache Disorders; Headache; Tension-Type Headache; Migraine Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cerebrospinal Fluid and Blood are collected and stored for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Episodic Headache: Participants experiencing headache of any type more than twice per year but less than 15 days per month. No interventions
- Chronic Headache: Participants experiencing headache more than 15 days per month for at least three consecutive months. No interventions
- Control: Participants reporting fewer than two headaches per year. No interventions

SUMMARY:
Study is aimed at determining why some patients with episodic headache proceed to chronic daily or near daily headaches. The Investigators seek to discover differences in brain anatomy and function, composition of cerebrospinal fluid, blood products, genetics, and patient phenotypes that might help explain this process.

DETAILED DESCRIPTION:
The purpose of our study is to better understand disease processes and risk factors involved in onset of chronic daily headaches/Chronic Migraines. Further, The Investigators hopes to learn more about the etiology and disease mechanisms to optimize treatment strategies and determine prophylactic measures.

Participation in this research study, will include online questionnaires, a blood sample, a lumbar puncture, and a magnetic resonance imaging (MRI) scan without contrast to measure brain activity. Participant may select to participate in a magnetic resonance imaging (MRI) scan and/ or lumbar puncture. participating in atleast 3 procedures is required (blood draw, online questionnaires , MRI and/or Spinal Tap.

The study recruits participants with headache ( any type of headaches), and patients with no headaches ( or less than 2/year). Participants do not need to have a specified headache type. All participants are asked to complete an on-line survey to characterize a number of phenotypic features felt to be relevant by the Investigators. Three independent study groups (imaging, proteomics/genetics, and phenotyping) analyze data independently and stratify the data. Then, by group analysis, correlation among the different modalities is sought to identify features that distinguish common elements that might help elucidate features that could predict which patients with episodic headache are likely to progress to chronic, and which patients without headache might be at greater risk to develop new daily persistent headache.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must agree to sign informed consent.
* Subject must be able to or at least with some help willing to complete online questionnaires in English .
* Willing to comply with study instructions.
* must speak and understand English

Exclusion Criteria:

*Any neurological condition, at the discretion of the Principal Investigator (PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anybody above 18 years of age regardless of their race, gender will be able to participate in this study.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2014-12-12 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of chronification of headache | five years
  Brain Imaging, Phenotyping and Proteomics data will be combined to learn headache mechanisms.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cowan, MD, FAAN, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woldeamanuel YW, Sanjanwala BM, Cowan RP. Deep and unbiased proteomics, pathway enrichment analysis, and protein-protein interaction of biomarker signatures in migraine. Ther Adv Chronic Dis. 2024 Sep 18;15:20406223241274302. doi: 10.1177/20406223241274302. eCollection 2024. PMID 39314676